CLINICAL TRIAL: NCT01397279
Title: Assessment of Liver Glucose Metabolism in Diabetic Subjects
Acronym: CLAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CLAVA
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Newly Diagnosed Type 2 Diabetes (During the Last 12 Months)
Keywords: type 2 diabetes; insulin sensitivity; hyperinsulinemic euglycemic clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botnia clamp (Active Comparator): hyperinsulinemic euglycemic clamp following intravenous glucose tolerance test
  Interventions: Biological: intravenous glucose tolerance test; Biological: hyperinsulinemic euglycemic clamp
- hyperinsulinemic euglycemic clamp (Active Comparator): hyperinsulinemic euglycemic clamp without previous intravenous glucose tolerance test
  Interventions: Biological: hyperinsulinemic euglycemic clamp

INTERVENTIONS:
Biological: intravenous glucose tolerance test — Administration of a 30% weight-adapted glucose bolus intravenously.
  Other Names: ivGTT
  Arms: Botnia clamp
Biological: hyperinsulinemic euglycemic clamp — Intravenous administration of 20% glucose and insulin over 3 hours
  Other Names: HEC

SUMMARY:
Type 2 diabetes is associated with hepatic insulin resistance. One consequence of insulin resistance of the liver is an altered hepatic glucose metabolism. This study investigates whether the whole body (M-value) and hepatic insulin sensitivity obtained by hyperinsulinemic euglycemic clamp is influenced by a preceding intravenous glucose tolerance test (Botnia Clamp) in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
The hyperinsulinemic euglycemic clamp represents the gold standard for measuring peripheral insulin sensitivity. The insulin sensitivity is described by the M-value,which is calculated from glucose infusion rates during the last 30min of the clamp.

Glucose is metabolised in the periphery: 50% by neural tissues, 20% by splanchnic bed and liver, 15% by skeletal muscle, 5% by adipose tissue and 10% by blood cells and other tissues. Under hyperinsulinemic conditions there is a strong shift in glucose utilization: 85% skeletal muscle and 15% by neural tissues, splanchnic bed and liver, adipose tissue, blood cells and other tissues. The contribution of skeletal muscle varies with different insulin sensitivity.

We now want to investigate whether there is a difference in tissue-specific insulin sensitivity measured from a Botnia clamp (intravenous glucose tolerance test (ivGTT) and following clamp) and a single hyperinsulinemic euglycemic clamp? After a 60min ivGTT blood glucose levels in type 2 diabetic subjects are still elevated compared to baseline. High blood glucose levels can influence several parameters and may also affect insulin sensitivity. Until now, it is not proven, that the clamp preceding ivGTT does not have a significant influence on the M-value.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetes (during the last 12 months)or non-diabetic subjects

Exclusion Criteria:

* severe chronic diseases
* hepatitis B, C oder HIV infection
* malignancies
* immune suppressive therapy
* psychiatric illnesses
* drug or alcohol abuse
* anemia
* renal dysfunction

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
M Value in hyperinsulinemic euglycemic clamp | 3h
  measurement of whole body insulin sensitivity with hyperinsulinamic euglicamic clamp

SECONDARY OUTCOMES:
Insulin-suppressed endogenous glucose production (liver insulin sensitivity) | 3h
  Insulin-suppressed endogenous glucose production (liver insulin sensitivity)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Study Director — Director German Diabetes Center; Michael Roden, Prof., MD, Principal Investigator — Director German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Kahl S, Nowotny B, Piepel S, Nowotny PJ, Strassburger K, Herder C, Pacini G, Roden M. Estimates of insulin sensitivity from the intravenous-glucose-modified-clamp test depend on suppression of lipolysis in type 2 diabetes: a randomised controlled trial. Diabetologia. 2014 Oct;57(10):2094-102. doi: 10.1007/s00125-014-3328-3. Epub 2014 Jul 22. PMID 25047649